CLINICAL TRIAL: NCT00860431
Title: K-STAR (Kremezin STudy Against Renal Disease Progression in Korea) Randomized, Open-label, Controlled Study
Brief Title: Kremezin Study Against Renal Disease Progression in Korea
Acronym: K-STAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: HK inno.N Corporation (Industry); Kureha Corporation (Industry)
Responsible Party: Yon Su Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-2008-355-0
Record Dates: First submitted 2009-03-09; First posted 2009-03-12 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — AST 120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Standard-of-care (conservative treatment)
- 2 (Experimental): AST-120 6g/day (3 times a day)
  Interventions: Drug: AST-120

INTERVENTIONS:
Drug: AST-120 — 6g/day (3 times a day)
  Arms: 2

SUMMARY:
1. To evaluate the effectiveness of AST-120 (spherical carbon adsorbent) added to standard-of-care therapy in moderate to severe Chronic Kidney Disease (CKD III-IV), on time to first occurrence of any event of the triple composite outcome of initiation of renal replacement therapy, decline of eGFR 50% or more or doubling of serum creatinine (sCr) when compared with standard-of-care group;
2. To evaluate the effectiveness of AST-120 (spherical carbon adsorbent) to GFR and proteinuria;
3. To evaluate the effectiveness of AST-120 (spherical carbon adsorbent) to health related quality of life;
4. To evaluate the safety and tolerability of long-term AST-120 therapy in patients with CKD;
5. To evaluate the all-cause mortality and hospitalization apart from those planned for operation and intervention)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 18 years or older
* CKD stage 3,4 (estimated GFR by Cockcroft-Gault equation 15-59 mL/min/1.73m^2)
* Followed up by responsible nephrologists more than 6 months
* eGFR checked 2 times or more during screening period
* eGFR declined or expected to decline >= 5mL/min/year or >=2.5mL/min/6 months
* Blood pressure <= 160/100 mmHg
* Blood pressure checked 3 times or more during screening period
* No significant change of medication for CKD

Exclusion Criteria:

* Patients who took medicine AST-120 or ketosteril within 2 months
* Received any investigational agent or participated in a clinical study within the previous 2 months
* History of gastrointestinal disease (active gastric ulcer, inflammatory bowel disease, hiatal hernia, or severe GI dysmotility)
* obstructive urologic disease and other reversible kidney diseases
* chronic kidney disease due to autosomal dominant polycystic kidney disease, ADPKD
* severe nephrotic syndrome, 10g or more/day(or random urine pCR >= 10.0)
* History of previous kidney transplant
* Heart failure (NYHA III-IV), uncontrolled arrhythmia, unstable angina
* Liver cirrhosis (Child-Pugh B,C)
* active infection, uncontrolled inflammatory disease
* progressive malignant disease
* cerebral infarction and intracranial hemorrhage within 6 months,except transient ischemic attack (TIA)
* uncontrolled blood sugar (HbA1c >10%)
* severe anemia, Hb <7g/dL
* Life expectancy less than 12 months at the point of randomization
* Pregnant and willing to bear child during study
* patients, inappropriate to study (researchers decided)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The development of a component of a triple composite endpoint (doubling of serum Cr, decline of estimated GFR 50% or more by C-G equation, initiation of renal replacement therapy) | approximately 49 months (at least 12 months for enrollment and 36 months for intervention, 1month for follow up)

SECONDARY OUTCOMES:
change of estimated GFR and urine protein excretion, Assessment of health related quality of life, all-cause mortality | approximately 49 months (at least 12 months for enrollment and 36 months for intervention, 1month for follow up)

CONTACTS AND LOCATIONS:
Overall Officials: Yon Su Kim, M.D.PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Baek SH, Cha RH, Kang SW, Park CW, Cha DR, Kim SG, Yoon SA, Kim S, Han SY, Park JH, Chang JH, Lim CS, Kim YS, Na KY. Circulating renalase predicts all-cause mortality and renal outcomes in patients with advanced chronic kidney disease. Korean J Intern Med. 2019 Jul;34(4):858-866. doi: 10.3904/kjim.2017.058. Epub 2017 Nov 29. PMID 29172403
- [Derived] Lee SW, Kim S, Na KY, Cha RH, Kang SW, Park CW, Cha DR, Kim SG, Yoon SA, Han SY, Park JH, Chang JH, Lim CS, Kim YS. Serum Anion Gap Predicts All-Cause Mortality in Patients with Advanced Chronic Kidney Disease: A Retrospective Analysis of a Randomized Controlled Study. PLoS One. 2016 Jun 1;11(6):e0156381. doi: 10.1371/journal.pone.0156381. eCollection 2016. PMID 27249416